CLINICAL TRIAL: NCT06159933
Title: Early Prone Positioning as a Rescue Therapy for Severe Primary Graft Dysfunction After Bilateral Lung Transplant.
Brief Title: Primary Graft Dysfunction, Pronation, Bilateral Lung Transplants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Annalisa Boscolo, Doctor, University of Padova
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: reference 4539/AO/18
Record Dates: First submitted 2023-11-28; First posted 2023-12-07 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Lung Transplant; Primary Graft Dysfunction
Keywords: pronation, end-stage lung disease
MeSH Terms: conditions — Primary Graft Dysfunction

STUDY DESIGN:
Intervention Model Description: Historic cohort enrolled between January 2020 and December 2021; Prospective enrollment from January 2022 to April 2023. According to our local protocol, until December 2021, all patients developing PGD >1 after LT were monitored in supine position for at least 24 hours, aiming at optimizing mechanical ventilation settings and right ventricular function, before considering PP. Only in case of radiological worsening or reduction in PaO2/FiO2 ratio patients were turned prone, generally between 24 and 48 hours after the diagnosis ('late PP' group), otherwise they were maintained supine ('supine' group). On the contrary, starting from January 2022 our local protocol was updated and all LT recipients developing PGD >1 were routinely turned prone within 24 hours after the diagnosis ('early PP').Patients were placed in PP for at least 16 hours before being turned back to the supine position when meeting predefined criteria previously published by Guèrin et al.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Historic cohort (SUPINE POSITIONING) (Experimental): According to our local protocol, until December 2021, all patients developing PGD >1 after LT were monitored in supine position for at least 24 hours, aiming at optimizing mechanical ventilation settings and right ventricular function, before considering PP. Only in case of radiological worsening or reduction in PaO2/FiO2 ratio patients were turned prone, generally between 24 and 48 hours after the diagnosis ('late PP' group), otherwise they were maintained supine ('supine' group).
  Interventions: Procedure: Supine positioning
- Historic cohort (LATE PRONATION) (Experimental): According to our local protocol, until December 2021, all patients developing PGD >1 after LT were monitored in supine position for at least 24 hours, aiming at optimizing mechanical ventilation settings and right ventricular function, before considering PP. Only in case of radiological worsening or reduction in PaO2/FiO2 ratio patients were turned prone, generally between 24 and 48 hours after the diagnosis ('late PP' group), otherwise they were maintained supine ('supine' group).
  Interventions: Procedure: Late pronation
- Prospective cohort (EARLY PRONATION) (Experimental): On the contrary, starting from January 2022 our local protocol was updated and all LT recipients developing PGD >1 were routinely turned prone within 24 hours after the diagnosis ('early PP').Patients were placed in PP for at least 16 hours before being turned back to the supine position when meeting predefined criteria previously published by Guèrin et al
  Interventions: Procedure: Early pronation

INTERVENTIONS:
Procedure: Supine positioning — According to our local protocol, until December 2021, all patients developing PGD >1 after LT were monitored in supine position for at least 24 hours, aiming at optimizing mechanical ventilation settings and right ventricular function, before considering PP. Only in case of radiological worsening or reduction in PaO2/FiO2 ratio patients were turned prone, generally between 24 and 48 hours after the diagnosis ('late PP' group), otherwise they were maintained supine ('supine' group).
  Arms: Historic cohort (SUPINE POSITIONING)
Procedure: Early pronation — According to our local protocol, starting from January 2022, all patients developing PGD >1 after LT were monitored in supine position for at least 24 hours, aiming at optimizing mechanical ventilation settings and right ventricular function, before considering PP. Only in case of radiological worsening or reduction in PaO2/FiO2 ratio patients were turned prone, generally between 24 and 48 hours after the diagnosis ('late PP' group), otherwise they were maintained supine ('supine' group).
  Arms: Prospective cohort (EARLY PRONATION)
Procedure: Late pronation — According to our local protocol, until December 2021, all patients developing PGD >1 after LT were monitored in supine position for at least 24 hours, aiming at optimizing mechanical ventilation settings and right ventricular function, before considering PP. Only in case of radiological worsening or reduction in PaO2/FiO2 ratio patients were turned prone, generally between 24 and 48 hours after the diagnosis ('late PP' group), otherwise they were maintained supine ('supine' group).
  Arms: Historic cohort (LATE PRONATION)

SUMMARY:
Proning manoeuvre as an early treatment for acute severe hypoxic respiratory failure has been implemented recently during the COVID-19 pandemic. This method was proposed more than fifty years ago to improve gas exchange : Proning Severe ARDS (PROSEVA) trial, however, was the milestone which demonstrated mortality benefit in patients with severe ARDS. Nevertheless, few analysis were performed on the effects of the prone position after lung transplantion (LT). The aim of the study is therefore to relate LT primary graft dysfunction (PGD) pathophysiology, which occurs in postoperative setting, to prone-positioning effects on ventilation-perfusion matching, improved lung compliance and clinical outcomes of impairedorgan patients.

DETAILED DESCRIPTION:
Lung transplant is the final stage of intervention in dramatic respiratory failure unresponsive to other medical or surgical treatments: reduced disability, improved life quality and extended life are outweighed by still high mortality and morbidity of LT, compared to other solid organs transplants. LT patient survival is undermined, above all, by PGD onset up to 72h in postoperative scenario. Acute lung injury, characterized by reperfusion and ischemia damage, evolves in pulmonary edema and severely inflammed graft status. Tipical radiological findings are bilateral spreading infiltrates, whose treatment was until some years ago mainly supportive, i.e. protective mechanical ventilation and fluid restriction. Two retrospective studies recently demonstrated favorable oxygenation response in terms of PaO2/fraction-of-inspired-oxygen (FiO2) ratio and lung compliance. Our purpose was to broaden gas-exchange results by the analysis of short-term outcomes (i.e duration of mechanical ventilation, reintubation or tracheostomy, anastomotical complications, organ rejection in 30 days, acute kindney injury development and/or filtration necessity, hospital length and mortality). Our aim is to assess through this pilot study if early pronation (realized within 24 hours from admission) has a more favorable outcome on patients developing moderate/severe PGD within the first 24 postoperative hours.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 y.o.
* First bilateral lung transplant
* PGD grade 2 or 3 within 24 hours from ICU admission Admission to ICU for post-operative monitoring after LTx
* Written informed consent obtained

Exclusion Criteria:

* Age < 18 years old
* PGD<2
* Single transplant
* Re-transplant
* IMV, venous-venous (V-V) or venous-arterial (V-A) extracorporeal membrane oxygenation (ECMO) before surgery
* Contraindications to prone positioning
* Refusal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
28-day ventilator free days | From ICU admission up to 28 post-operative days (POD)
  Days free from invasive mechanical ventilation after lung transplant

SECONDARY OUTCOMES:
Invasive mechanical ventilation (IMV) | From ICU adminission up to liberation from invasive mechanical ventilation
  Duration of IMV
Blood gas exchanges (PaO2 /FiO2 PaCo2, pH) | Within 24hours from ICU admission, at 72 hours later, in supine and prone position
  Emogas analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Università Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No